CLINICAL TRIAL: NCT04019899
Title: Effects of Supplementation With Myo-inositol, Vitamin D3, Folic Acid and Melatonin on IVF Outcomes
Brief Title: Myo-inositol and Vitamin D3 During IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000153
Record Dates: First submitted 2019-07-10; First posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Female Infertility
MeSH Terms: conditions — Infertility, Female | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator)
  Interventions: Dietary Supplement: control group
- Study group (Experimental)
  Interventions: Dietary Supplement: study group

INTERVENTIONS:
Dietary Supplement: control group — * 2 g Myo-Inositol, 50 mg Alpha-Lactalbumin and 200 µg folic acid (1 sachet/day in the morning): from the first day of the menstrual cycle until 14 days after embryo transfer. If pregnancy occurs, until the 12th week of gestation.
  * 600 mg Myo-Inositol, 200 µg folic acid, 1 mg melatonin (1 soft capsule/day in the evening): from the first day of the menstrual cycle until hCG administration. If pregnancy occurs, until the 12th week of gestation.
  Arms: Control group
Dietary Supplement: study group — * 2 g Myo-Inositol, 50 mg Alpha-Lactalbumin and 200 µg folic acid (1 sachet/day in the morning): from the first day of the menstrual cycle until 14 days after embryo transfer. If pregnancy occurs, until the 12th week of gestation.
  * 600 mg Myo-Inositol, 200 µg folic acid, 1 mg melatonin (1 soft capsule/day in the evening): from the first day of the menstrual cycle until hCG administration;
  * 600 mg Myo-Inositol, 200 µg folic acid, 1 mg melatonin, 50 µg vitamin D3 as cholecalciferol (1 soft capsule/day in the evening) substitutes the previous treatment at hCG administration and lasted until 14 days after embryo transfer. If pregnancy occurs, until the 12th week of gestation.
  Arms: Study group

SUMMARY:
Administration of a multicomponent dietary supplement (myo-inositol, vitamin D3, folic acid and melatonin) to women undergoing IVF procedures.

The aim of the study is to monitor the effects on the pregnancy, implantation and abortion rates.

ELIGIBILITY:
Inclusion Criteria:

* BMI (kg/m2): 18.5 - 24.9
* basal FSH on day 3 <15 mIU/ml

Exclusion Criteria:

* presence of insulin resistance (IR)
* hyperglycaemia, hyperprolactinemia, hypothyroidism or androgen excess
* diagnosis of PCOS (according to Rotterdam ESHRE-ASRM Sponsored PCOS consensus workshop group)
* intake of hormones or drugs that can potentially influence the ovulation
* FSH>15 on day 3

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Implantation rate | Single time-point: at 6 weeks of pregnancy
  number of gestational sacs observed at ecographic screening divided by the number of embryos transferred
oocyte and embryo quality | Single time-point: respectively, 12 days and 15 days after the beginning of Controlled Ovarian Hyperstimulation
  Classification of the morphological aspects under the optical microscope
clinical pregnancy | Single time-point: at 14 days from embryo transfer
  Positive beta-hCG test after embryo transfer

SECONDARY OUTCOMES:
Gemellarity | Single time-point: at 6 weeks of pregnancy
  Multiple gestational sacs observed at ecographic screening
Abortion rate | Single time-point: at 6 weeks of pregnancy
  Loss of pregnancy
Number of FSH IU used for controlled ovarian hyperstimulation | Single time-point: about 10 days after the beginning of Controlled Ovarian Hyperstimulation
  Ovarian ultrasound investigation and serum estradiol level

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Alma Res, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No